CLINICAL TRIAL: NCT01341080
Title: Varenicline for the Treatment of Postural and Gait Dysfunction in Parkinson Disease
Brief Title: Varenicline for Gait and Balance Impairment in Parkinson Disease
Acronym: Chantix-PD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Principal Investigator, Deborah Hall, MD, MD, Rush University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WS813511
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Results first posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Parkinson Disease
Keywords: Balance; Postural impairment; Falls; Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Varenicline; Sugars

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Varenicline (Experimental)
  Interventions: Drug: Varenicline
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Sugar pill

INTERVENTIONS:
Drug: Varenicline — Varenicline 1mg twice daily for eight weeks after a one week dose escalation period.
  Other Names: Chantix
  Arms: Varenicline
Drug: Sugar pill — 1mg twice daily for eight weeks after a one week dose escalation phase.
  Arms: Sugar pill

SUMMARY:
The purpose of this study is to determine if varenicline is effective in improving gait and balance impairment in patients with Parkinson disease.

DETAILED DESCRIPTION:
Parkinson disease (PD) is a clinical entity characterized by bradykinesia, rigidity, tremor, and postural instability. Current treatments primarily focus on replacement of dopamine to compensate for the degeneration of the substantia nigra pars compacta dopaminergic neuronal population. Though dopamine treats many of the motor symptoms of PD, postural instability (which often leads to falls) typically is least responsive to therapy. More recently, the degeneration of the cholinergic system arising from the pedunculopontine nucleus (PPN) in the brainstem has been implicated in gait dysfunction in PD. Striatal cholinergic inputs are supplied from the PPN both via the intralaminar complex of the thalamus and through direct inputs. The primary subtypes of cholinergic receptors present in the striatum are nicotinic and include α4β2, α6β2, and α7 receptors. Varenicline (Chantix) is a novel partial α4β2 agonist and full α7 agonist developed as an aid for smoking cessation and has been shown in initial studies to improve imbalance in patients with inherited spinocerebellar ataxia. The unique method of action of varenicline may make it an ideal drug for the treatment of balance impairment in PD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be diagnosed with Parkinson Disease (PD) by the United Kingdom (UK) Brain Bank criteria.
* Subjects will have to be at least stage 2 on the Hoehn and Yahr staging system of PD and have a history of at least 1 fall or near fall in the last 6 months
* Subjects must have a stable medication regimen.
* All subjects will be over the age of 40 in an attempt to exclude inherited forms of parkinsonism.
* Serum creatine kinase, complete metabolic panel, complete blood count, liver function tests, renal function tests, platelets and EKG are within normal limits (results obtained from primary care physician and dated within the past 6 months or obtained at screening visit).

Exclusion Criteria:

* Hoehn and Yahr stage V subjects.
* Subjects with a history of major psychiatric disorder, deep brain stimulation surgery, recent cerebral trauma, cardiac arrhythmia, or renal insufficiency.
* A cardiovascular procedure in the last 5 years (eg, percutaneous transluminal coronary angioplasty) or have cardiovascular instability (including myocardial infarction or unstable angina). Other cardiovascular exclusions include uncontrolled hypertension, significant neurological sequelae of cerebrovascular disease, peripheral vascular disease with prior amputation, or severe congestive heart failure (New York Heart Association class III or IV).
* Concurrent treatment with any monoamine oxidase inhibitors (MAOIs), bupropion (Wellbutrin), or nicotine patches.
* Dementia or other psychiatric illness that prevents the patient from giving informed consent (Folstein Mini Mental Status Exam score less than 25).
* Concurrent treatment with trihexyphenidyl (Artane) or benztropine mesylate (Cogentin).
* Significant degree of dysphagia, by history.
* Legal incapacity or limited legal capacity.
* Presence of severe renal disease (BUN 50% greater than normal or creatinine clearance <60 mL/min) or hepatic disease.
* Abnormal creatine kinase and/or platelet count in the past 6 months (as determined by lab reports obtained from primary care physicians or conducted at baseline).
* Use of varenicline within the previous 30 days.
* Women of childbearing potential who are pregnant at the time of screening or who will not use adequate protection during participation of the study.
* Allergy/sensitivity to the drug or its formulations.
* Concurrent participation in another clinical study.
* Active substance or tobacco use or dependence.
* Moderate or severe chronic obstructive pulmonary disease.
* Serious illness (requiring systemic treatment/or hospitalization) until the subject either completes therapy or is clinically stable on therapy, in the opinion of the site investigator, for at least 60 days prior to study entry.
* Inability or unwillingness of the subject or legal guardian/representative to give written informed consent.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12-28 (Actual); Primary Completion 2018-11-02 (Actual); Study Completion 2018-11-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah A Hall, MD, PhD, Principal Investigator — Rush University Medical Center
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] Bohnen NI, Muller ML, Koeppe RA, Studenski SA, Kilbourn MA, Frey KA, Albin RL. History of falls in Parkinson disease is associated with reduced cholinergic activity. Neurology. 2009 Nov 17;73(20):1670-6. doi: 10.1212/WNL.0b013e3181c1ded6. PMID 19917989
- [Background] Qutubuddin AA, Pegg PO, Cifu DX, Brown R, McNamee S, Carne W. Validating the Berg Balance Scale for patients with Parkinson's disease: a key to rehabilitation evaluation. Arch Phys Med Rehabil. 2005 Apr;86(4):789-92. doi: 10.1016/j.apmr.2004.11.005. PMID 15827933
- [Background] Zesiewicz TA, Sullivan KL. Treatment of ataxia and imbalance with varenicline (chantix): report of 2 patients with spinocerebellar ataxia (types 3 and 14). Clin Neuropharmacol. 2008 Nov-Dec;31(6):363-5. doi: 10.1097/WNF.0b013e31818736a9. PMID 19050414
- [Background] Perez XA, Quik M. Focus on alpha4beta2* and alpha6beta2* nAChRs for Parkinson's Disease Therapeutics. Mol Cell Pharmacol. 2011;3(1):1-6. PMID 21499569
- [Background] Bohnen NI, Albin RL. The cholinergic system and Parkinson disease. Behav Brain Res. 2011 Aug 10;221(2):564-73. doi: 10.1016/j.bbr.2009.12.048. Epub 2010 Jan 7. PMID 20060022
- [Background] Karachi C, Grabli D, Bernard FA, Tande D, Wattiez N, Belaid H, Bardinet E, Prigent A, Nothacker HP, Hunot S, Hartmann A, Lehericy S, Hirsch EC, Francois C. Cholinergic mesencephalic neurons are involved in gait and postural disorders in Parkinson disease. J Clin Invest. 2010 Aug;120(8):2745-54. doi: 10.1172/JCI42642. Epub 2010 Jul 12. PMID 20628197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruitment from the Parkinson's Disease and Movement Disorder clinic at Rush University Medical Center over the course of the study (2011-2018).
Pre-assignment Details: 40 participants signed an informed consent form and 36 were randomized. Six participants terminated participation early, with 2 having sufficient data for last observations carried forward intention-to-treat analyses. The remaining 32 were used in the analysis.
Period: Overall Study
Arm/Group | Varenicline | Sugar Pill
Started | 18 (Subjects were randomly assigned to Varenicline) | 18 (Subjects were randomly assigned to placebo)
Completed | 15 (Completed) | 17 (Completed)
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Population: 36 participants were randomized. Six participants terminated participation early with 2 having sufficient data for last observations carried forward. 32 were used in the analysis and demographics are reported here.
Groups:
- Total: Total of all reporting groups
Arm/Group | Varenicline | Sugar Pill | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants] — Population: Forty participants signed an informed consent form and 36 were randomized. Six participants terminated participation early, with 2 having sufficient data for last observations carried forward intention-to-treat analyses. The remaining sample was 32 participants.Fifteen participants were randomized to receive varenicline and 17 to placebo.
  Participants
    number analyzed (Participants) | 15 | 17 | 32
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 3 | 3 | 6
    >=65 years | 12 | 14 | 26
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Forty participants signed an informed consent form and 36 were randomized. Six participants terminated participation early, with 2 having sufficient data for last observations carried forward intention-to-treat analyses. The remaining sample was 32 participants.Fifteen participants were randomized to receive varenicline and 17 to placebo.
  years
    number analyzed (Participants) | 15 | 17 | 32
    (all) | 71.93 (8.5) | 70.24 (7.9) | 71.03 (8.134)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Forty participants signed an informed consent form and 36 were randomized. Six participants terminated participation early, with 2 having sufficient data for last observations carried forward intention-to-treat analyses. The remaining sample was 32 participants.Fifteen participants were randomized to receive varenicline and 17 to placebo.
  Participants
    number analyzed (Participants) | 15 | 17 | 32
    Female | 3 | 3 | 6
    Male | 12 | 14 | 26
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: 36 participants were randomized and six participants terminated early. 2 had sufficient data for last observations carried forward. The remaining sample of 32 was used in the analysis.
  Participants
    White: number analyzed (Participants) | 15 | 17 | 32
    White | 15 | 17 | 32
Region of Enrollment [Number; unit: participants] — Population: Forty participants signed an informed consent form and 36 were randomized. Six participants terminated participation early, with 2 having sufficient data for last observations carried forward intention-to-treat analyses. The remaining sample was 32 participants.Fifteen participants were randomized to receive varenicline and 17 to placebo.
  participants
    United States: number analyzed (Participants) | 15 | 17 | 32
    United States | 15 | 17 | 32
Unified Parkinson's Disease Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The UPDRS part III measures motor signs of Parkinson's disease. The maximum Part III score is 108 and the minimum is 0. The higher the score, the worse the motor findings.
  units on a scale | 33.1 (9.7) | 35.7 (12.7) | 34.74 (11.558)

OUTCOME MEASURES:

1. Primary Outcome: Berg Balance Scale
Description: Efficacy was measured as a change on the Berg Balance Scale (BBS) from baseline to the end of the study after 8 weeks on drug. The BBS is a 14-item measure consisting of basic balance tasks, with a final score indicative of overall balance ability. The maximum score is 56 and minimum is 0. Higher scores reflect better balance.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Sugar Pill
Number analyzed (Participants) | 15 | 17
score on a scale
  Baseline | 43.93 (1.97) | 41.14 (2.55)
  End Point | 43.25 (1.84) | 45.13 (2.34)
Statistical Analysis 1: Comparison: Varenicline vs Sugar Pill; Efficacy was measured as a change on the Berg Balance Scale (BBS) from baseline to the end of study after 8 weeks on drug. The BBS has a scale range of 0-56, with 56 indicating normal balance. To evaluate efficacy, repeated measures analysis of variance was run on BBS scores. The scale score was the dependent measure, time point (baseline or end of study) was the repeat measure, and treatment group (varenicline or sugar pill) was the independent measure. Significance was defined as alpha <0.05; Test type: Other; p = 0.05, Repeated measures analysis or variance; Cohen's d = 0.15, 95% CI 2-sided [-4.01 to 4.61]

2. Secondary Outcome: Frontal Assessment Battery
Description: The change in cognitive functioning was measured with the Frontal Assessment Battery (FAB, score range 0-18) and the Mini-Mental State Exam (MMSE, score range 0-30) from baseline to 8 weeks on drug. High scores on both scales indicate better performance. The FAB measures executive functioning and consists of the following 6 sections: conceptualization, mental flexibility, motor programming, sensitivity to interference, inhibitory control, and environmental autonomy.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Sugar Pill
Number analyzed (Participants) | 15 | 17
score on a scale
  Baseline | 17.40 (0.97) | 15.25 (2.77)
  End point | 17.70 (2.16) | 15.19 (2.74)
Statistical Analysis 1: Comparison: Varenicline vs Sugar Pill; Change in cognitive functioning was measured in part with the Frontal Assessment Battery (FAB) from Baseline to 8 weeks on drug. Repeated analysis of variance was run on the FAB scores. Scale cores was the dependent measure, time point (Baseline or end of study) was the repeated measure, and treatment group (varenicline or sugar pill) was the independent measure. Significant was defined as <0.05; Test type: Other; p = 0.05, Repeated measures analysis or variance; Cohen's d = 0.16, 95% CI 2-sided [-1.39 to 1.53]

3. Secondary Outcome: Mini Mental Status Exam (MMSE)
Description: The change in cognitive functioning was measured with the Mini-Mental State Exam (MMSE) from baseline to 8 weeks on drug. The maximum score on the MMSE is 30 and lowest score 0, with higher score indicating better cognitive function.
Time Frame: 9 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Varenicline | Sugar Pill
Number analyzed (Participants) | 15 | 17
score on a scale
  Baseline | 29.08 (1.17) | 28.19 (1.72)
  End point | 28.00 (2.00) | 28.13 (1.7)
Statistical Analysis 1: Comparison: Varenicline vs Sugar Pill; Change in cognitive functioning was measured in part with the Mini Mental State Exam (MMSE) from Baseline to 8 weeks on drug. Repeated analysis of variance was run on the MMSE scores. Scale score was the dependent measure, time point (Baseline or end of study) was the repeated measure, and treatment group (varenicline or sugar pill) was the independent measure. Significant was defined as <0.05; Test type: Other; p = 0.05, Repeated measures analysis or variance; Cohen's d = 0.81, 95% CI 2-sided [-0.40 to 1.40]

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout subject participation (e.g. 9 weeks).
Description: Definition: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research. During follow-up visits and phone calls subjects were asked if they had experienced any problems and/or side effects since their last visit.
Arm/Group | Varenicline | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

LIMITATIONS AND CAVEATS:
The sensitivity of the BBS is poor to moderate, with frequent uncertainty in its scoring; The study also faced challenges in recruitment, which was slow and spanned 8 years, potentially biasing the sample; High attrition resulted in a smaller sample size than estimated by power analysis; Although the authors intended to recruit tremor predominant and PIGD patients in equal numbers, the PIGD subtype was overrepresented. Thus, the PIGD subtype was unintentionally favored.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2011-08-23): https://cdn.clinicaltrials.gov/large-docs/80/NCT01341080/Prot_SAP_000.pdf
  • Informed Consent Form (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT01341080/ICF_001.pdf